CLINICAL TRIAL: NCT03264222
Title: Safety of a New Security Device in Patients With Implanted Cardiac Electronic Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Bayerisches Staatsministerium für Wirtschaft (Unknown); R & S GmbH und Co KG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GER-EP-017
Record Dates: First submitted 2017-06-26; First posted 2017-08-29 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Electromagnetic Interference

STUDY DESIGN:
Intervention Model Description: Prospective cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposition to safety screening (Other): One armed study with exposition to a new safety device (model QPS100) using radiofrequency technology
  Interventions: Other: Security screening procedure

INTERVENTIONS:
Other: Security screening procedure — Screening procedure with security device (model QPS 100)

SUMMARY:
Patients with implantable cardiac electronic devices will be exposed to a new safety device and evaluated for potential electromagnetic interference.

DETAILED DESCRIPTION:
Patients with implanted pacemakers or defibrillators will undergo a screening procedure with an innovative security device. Evaluation will be made with respect to the occurrence of interference.

ELIGIBILITY:
Inclusion Criteria:

* implantable pacemaker or defibrillator in situ

Exclusion Criteria:

* malfunction of implantable pacemaker or defibrillator
* low battery voltage of implanted cardiac electronic device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Electromagnetic interference | 10 minutes
  Occurrence of electromagnetic interference

CONTACTS AND LOCATIONS:
Overall Officials: Christof Kolb, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lennerz C, O'Connor MJ, Blazek P, Weigand S, Grebmer C, Reif S, Friedrich L, Reents T, Bourier F, Schunkert H, Deisenhofer I, Kolb C. Modern Security Screening and Electromagnetic Interference With Cardiac Implantable Electronic Devices. J Am Coll Cardiol. 2020 Mar 17;75(10):1238-1239. doi: 10.1016/j.jacc.2020.01.012. No abstract available. PMID 32164898